CLINICAL TRIAL: NCT01183910
Title: A Randomized, Double-Blind, Placebo-Controlled Study To Assess the Safety and Efficacy of a Novel Oral Natural Extract for the Treatment of Senile Purpura
Brief Title: A Novel Oral Natural Extract for the Treatment of Senile Purpura
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nexgen Dermatologics, Inc. (Industry)
Responsible Party: GARY BERLIN, ESQUIRE, NEXGEN DERMATOLOGICS, INC.
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 021775
Record Dates: First submitted 2010-08-16; First posted 2010-08-18 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: PURPURA
Keywords: PURPURA; SENILE PURPURA; BATEMAN'S PURPURA
MeSH Terms: conditions — Purpura | interventions — Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calcium carbonate placebo pill (Placebo Comparator): Placebo medication to treat the appearance of the skin in patients with senile purpura
  Interventions: Dietary Supplement: Calcium Carbonate
- Nutraceutical (Active Comparator): Patients take a novel, natural nutraceutical product to improve the appearance of the skin of patients with senile purpura
  Interventions: Dietary Supplement: Citrus Bioflavanoid Blend

INTERVENTIONS:
Dietary Supplement: Citrus Bioflavanoid Blend — Pill Taken Twice a Day
  Arms: Nutraceutical
Dietary Supplement: Calcium Carbonate — Oral Tablet Taken Twice a Day
  Arms: Calcium carbonate placebo pill

SUMMARY:
A randomized, double-blind, placebo controlled study to assess the safety and effectiveness of a novel oral natural extract to improve the appearance of the skin of patients with senile purpura.

ELIGIBILITY:
Inclusion Criteria:

* Patients with evidence of purpura on physical exam

Exclusion Criteria:

* Preexisting condition that would not allow the patients to take oral calcium supplement

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-07 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
IMPROVEMENT IN PATIENT'S SKIN APPEARANCE WITH SENILE PURPURA | 6 WEEKS

SECONDARY OUTCOMES:
ADVERSE EFFECTS IN PATIENTS WITH SENILE PURPURA TAKING THIS MEDICATION | 6 WEEKS

CONTACTS AND LOCATIONS:
Overall Officials: JOSHUA M BERLIN, MD, Principal Investigator — STUDY PROTOCOL, INC
Locations (1):
- Berlin Center of Medical Aesthetics, Boynton Beach, Florida, United States